CLINICAL TRIAL: NCT04953897
Title: A Phase 1b, Open-label, Parallel Group, Multiple-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Oral Decitabine and Cedazuridine (ASTX727) in Cancer Patients With Severe Renal Impairment and Cancer Patients With Normal Renal Function
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of Oral Decitabine and Cedazuridine in Cancer Patients With Renal Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTX727-17; 2024-516291-16-00 (EU CTIS Number)
Record Dates: First submitted 2021-06-30; First posted 2021-07-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: Severe Renal Impairment (Experimental): Cancer participants with severe renal impairment not requiring dialysis (creatinine clearance [CLcr] <30 mL/min/1.73m^2)
  Interventions: Drug: ASTX727
- Group B: Normal Renal Function (Active Comparator): Cancer participants with normal renal function (CLcr ≥80 mL/min/1.73m^2)
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: ASTX727 — Multiple-dose oral administration of once-daily decitabine (35 mg) and cedazuridine (100 mg)
  Other Names: Oral decitabine and cedazuridine

SUMMARY:
This is a Phase 1b, multicenter, open-label, PK, and safety study of multiple oral doses of oral decitabine and cedazuridine (formerly known as ASTX727) as a fixed-dose combination of decitabine 35 milligrams (mg) and cedazuridine 100 mg in cancer participants with severe renal impairment and cancer participants with normal renal function as matched control participants. Adult participants with acute myeloid lymphoma (AML), myelodysplastic syndrome (MDS), or solid tumors who are candidates to receive oral decitabine and cedazuridine will be enrolled in this study. Study duration per participant is approximately up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with the study procedures, understand the risks involved in the study, and provide legally effective informed consent before the first study-specific procedure; specifically able to comply with the PK assessment schedule during the first treatment cycle.
* Participants must have a histologically or cytologically confirmed malignancy as follows:

  1. A solid tumor that is metastatic or unresectable and for which standard life-prolonging measures are not available.

     or
  2. AML or MDS. or
  3. A hematologic malignancy other than AML or MDS for which standard life-prolonging measures are not available.
* For participants with AML/MDS only:

  1. Cytologically or histologically confirmed diagnosis of AML (except M3 acute promyelocytic leukemia) or MDS according to the 2008 World Health Organization (WHO) classification or
  2. Participants with frontline MDS or treatment naïve AML not suitable for induction therapy (e.g., age >75 years, Eastern Cooperative Oncology Group [ECOG] performance ≥2, severe pulmonary disorder, total bilirubin 1.5 × upper limit of normal [ULN]); or
  3. Platelet count ≥25,000/per microliter (μL); or
  4. Absolute neutrophil count (ANC) ≥100 cells/μL.
* For participants with only hematologic malignancies other than AML or MDS, or solid tumors:

  1. Platelet count ≥100,000/μL; and
  2. ANC ≥1000 cells/μL.
* ECOG performance status of 0 to 3.
* Adequate hepatic function defined as:

  1. Total or direct bilirubin ≤1.5X upper limit of normal (ULN); and
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5X ULN.
* Participants must have a body surface area (BSA)-adjusted CLcr using to the Cockcroft-Gault equation:

  1. Participants without renal impairment (Group B): ≥80 mL/min/1.73m^²;
  2. Participants with severe renal impairment (Group A): <30 mL/min/1.73m^², not requiring dialysis;
  3. CLcr must be stable with <30% deviation allowed from screening to Day -1 (Baseline). Participants shifting outside the prospected renal function category (normal renal function or severe renal function) on Day-1 Baseline need to be agreed by Taiho medical expert whether they are allowed to remain in the original category that was assessed at screening.
* No major surgery within 30 days of first administration of oral decitabine and cedazuridine.
* Life expectancy of at least 3 months.
* Women of childbearing potential (according to recommendations of the Clinical Trial Facilitation Group) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.
* Women of childbearing potential must agree to practice 1 highly effective contraceptive measure of birth control with low user dependency and must agree not to become pregnant for 6 months after completing treatment.
* Male participants with female partners of childbearing potential must agree to use a male condom and advise his partner to practice 1 highly effective contraceptive measure of birth control (user dependent or with low user dependency) and must agree not to father a child while receiving treatment with oral decitabine and cedazuridine for at least 3 months after completing treatment.

Exclusion Criteria:

* Treatment with azacitidine or decitabine within 4 weeks before Screening. Prior cytotoxic chemotherapy for AML except for hydroxyurea to control high white blood cell (WBC) counts.
* Hospitalization for more than 2 days for documented febrile neutropenia, pneumonia, sepsis, or systemic infection 30 days prior to first dose.
* Treatment with any investigational medicinal product (IMP), investigational therapy, chemotherapy, immunotherapy, or targeted therapy within 2 weeks or 5 half-lives, whichever is longer, before the first dose of study treatment, or ongoing clinically significant adverse events from previous treatment.
* Concurrent MDS therapies, including lenalidomide, cyclosporine/tacrolimus, granulocyte-colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor, etc. Prior treatment with these agents is permitted, provided that completion is at least 1 week before the first dose of study treatment. Short-term use of G-CSF for febrile neutropenia is permitted at the discretion of the treating physician and should be guided by accepted practice or institutional guidelines. Hematopoietic growth factors will not be routinely used unless cleared by Taiho medical expert.
* Administration of live (attenuated) vaccines within 4 weeks before the first administration of oral decitabine and cedazuridine until after the follow-up visit. Other vaccines, e.g., inactivated or ribonucleic acid (RNA)-based, may be administered but should not occur from 7 days before first administration of oral decitabine and cedazuridine until after the follow-up visit.
* High medical risk because of other conditions such as uncontrolled systemic diseases, active uncontrolled infections, or comorbidities that may put the participants at risk of not being able to complete 1 cycle of treatment.
* Conditions which likely promote delayed ventricular repolarization (QT prolongation):

  1. Corrected QT interval (QTc) using Fridericia's correction (QTcF) at Screening or Day -1 >470 milliseconds (ms) for males and >480 ms for females or
  2. History or disposition for torsades des pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT Syndrome) or
  3. Concomitant medications that prolong the QT/QTc interval
* Cardiac abnormalities or unstable cardiovascular conditions:

  1. Unstable ischemic heart disease or severe heart failure (New York Heart Association Class III or IV) or
  2. Uncontrolled treated/untreated hypertension (defined as a mean of 3 repeated measurements for systolic blood pressure ≥ 180 millimeters of mercury (mmHg) and/or diastolic blood pressure ≥ 110 mmHg; current or documented history of repeated clinically significant hypotension or severe episodes of orthostatic hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg).
* Known significant mental illness or other condition, such as active alcohol or other substance abuse or addiction, that in the opinion of the investigator predisposes the participants to high risk of noncompliance with the protocol.
* In participants with AML/MDS, rapidly progressive or highly proliferative disease or other criteria that render the participants at high risk of requiring intensive cytotoxic chemotherapy within the next 3 months.
* Life-threatening illness or severe organ system dysfunction, such as uncontrolled congestive heart failure or chronic obstructive pulmonary disease, or other reasons including laboratory abnormalities, that in the investigator opinion, could compromise the participant safety, interfere with the absorption or metabolism of oral decitabine and cedazuridine, or compromise completion of the study or integrity of the study outcomes.
* Untreated central nervous system (CNS) metastases. Participants with treated CNS metastases are eligible provided they have been clinically stable for at least 4 weeks before screening.
* Participants infected with human immunodeficiency virus (HIV).
* Participants with active hepatitis B or hepatitis C infection.
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
* Average intake of more than 24 units of alcohol per week for male participants and 17 units per week for female participants (1 unit of alcohol equals 10 milliliters (mL) of pure alcohol, i.e., approximately 250 mL of beer, 75 mL of wine or 25 mL of spirits).
* Donation or loss of more than 500 mL of blood within 60 days prior to the first study drug administration.
* Hypersensitivity to decitabine, cedazuridine, or any of the excipients in oral decitabine and cedazuridine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: 5-day Cumulative Area Under the Concentration-time Curve Within 1 Dosing Interval (AUCtau) | Predose and at multiple timepoints post-dose from Day 1 to Day 5
  AUCtau from Day 1 to Day 5 for decitabine.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter: Apparent Clearance (CL/F) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  CL/F of decitabine and cedazuridine.
Pharmacokinetic Parameter: Renal Clearance (CLR) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  CLR of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Apparent Nonrenal Clearance (CLNR/F) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  CLNR/F of decitabine and cedazuridine.
Pharmacokinetic Parameter: Time to Maximum Observed Plasma Concentration (Tmax) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  Tmax of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Maximum Observed Plasma Concentration (Cmax) | Predose and at multiple timepoints post-dose on Days 1, 2, and 5
  Cmax of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Plasma Concentration Prior to Dosing (Ctrough) | Predose on Days 2, 3, 4 and 5
  Ctrough of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Area Under the Concentration-time Curve from Time 0 (Time of Dosing) to Time t | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  AUCt of decitabine, cedazuridine, and cedazuridine-epimer, where t is the last time point with concentrations above the lower limit of quantitation.
Pharmacokinetic Parameter: AUC Within 1 Dosing Interval (AUCtau) | Predose on Day 1 to Day 2, Day 2 to Day 3, and Day 5 to Day 6 and at multiple timepoints on Day 1 to Day 2, Day 2 to Day 3, and Day 5 to Day 6
  AUCtau of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: AUC From Time 0 Extrapolated to Infinity (AUC0-inf) | Predose and at multiple timepoints post-dose on Days 1, 2, and 5
  AUC0-inf of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Terminal Elimination Phase Rate Constant (λz) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  λz of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Terminal Elimination Half-life (t1/2) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  t1/2 of decitabine, cedazuridine, and cedazuridine-epimer.
Pharmacokinetic Parameter: Apparent Volume of Distribution During Terminal Phase (Vz/F) | Predose from Day 1 to Day 5 and at multiple timepoints post-dose from Day 1 to Day 8
  Vz/F of decitabine and cedazuridine.
Pharmacokinetic Parameter: Fraction of Administered Drug Excreted into Urine (Fe/F) | Predose on Day 1 and at multiple timepoints post-dose from Day 1 to Day 6
  Fe/F of decitabine and cedazuridine.
Pharmacokinetic Parameter: Cumulative Amount Excreted from Time 0 to the Time of the Last Quantifiable Sample (Aelast) | Predose on Day 1 and at multiple timepoints post-dose from Day 1 to Day 6
  Aelast of decitabine, cedazuridine, and cedazuridine-epimer.
Safety Parameter: Number of Participants with Adverse Events (AEs) | Up to 8 weeks
  Adverse events included any untoward medical occurrence in a participant administered a drug; it does not necessarily have to have a causal relationship with this treatment also including clinically meaningful findings in laboratory safety tests, vital signs, physical examinations, and electrocardiogram (ECG) findings.

CONTACTS AND LOCATIONS:
Locations (21):
- MD Anderson, Houston, Texas, United States
- Armenia (4):
  - Erebuni Medical Center, Yerevan
  - Hematology Center After Prof. R. Yeolyan (Adult Blood Disorders), Yerevan
  - Hematology Center After Prof. R. Yeolyan (Clinic of Adults Oncology), Yerevan
  - National Center of Oncology Named After V.A. Fanarjyan, Yerevan
- Complex Oncology Center - Plovdiv - Base II, Plovdiv, Bulgaria
- BIO1, Vilnius, Lithuania
- Centrum Badań Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw, Poland
- Romania (2):
  - Institutul Oncologic Bucuresti - Prof. Dr. Alexandru Trestioreanu, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
- Summit Clinical Research s.r.o, Bratislava, Slovakia
- Spain (10):
  - START Barcelona - Hospital HM Nou Delfos, Barcelona
  - Hospital Universitari Dexeus - Grupo Quirónsalud, Barcelona
  - START Rioja - Hospital de San Pedro, La Rioja
  - Hospital Universitari Arnau de Vilanova, Lleida
  - START Madrid - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - START Madrid - CIOCC - HM Sanchinarro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca (Hematology Dept), Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca (Solid Tumor Dept), Murcia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No